CLINICAL TRIAL: NCT01433341
Title: Evaluation of Postural Control After Exercise in Athletes Using Tetra Axial Posturography (tetrax1)
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MeirMc06611TIL
Record Dates: First submitted 2011-09-12; First posted 2011-09-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: Normal young athletes

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Young athletes

SUMMARY:
Tetra-ataxiametric posturography is based on the measurement and computerized elaboration of electronic signals emitted by four footplates, one for each heel and toe, respectively. These are sensitive to vertical pressure produced by a subject standing straight but in various positions (feet parallel, in tandem, eyes closed, on pads, etc.). The method yields additional parameters not obtained by the traditional monoplate stabilometers, namely, weight-distribution patterns and correlation among six combinations of paired outputs from the two heels, two toes, heel/toe of each foot, and the two diagonals (tetra-ataxiametric synchronizations).

Most athletic injuries occur at the end of an activity, when the participant is fatigue. It is likely that significant portion of the injuries result from instability of the lower extremity joints as a consequence of fatigue of the stabilizing muscles. Muscle fatigue increase postural sway, impaired muscle control, and increase the onset delay of movement. Comparing pre-exercise with post-exercise results for each athlete, should detect significant and clinically meaningful differences with the Tetra-ataxiametric measures of stability, interaction between Fourier Spectral Power Ranges of body sway, weight distributions, and synchronizations of toe parts. The method is suitable for young subjects, and the equipment is portable and tests can be conveniently carried out in a child's familiar training setting and right before/after exercise.

The goal of the present study is to measure the balance of the athletes after different types of exercises, to measure the ability of the athletes to recover different types of exercises, and to measure the influence of increasing physical fitness on balance ability. Fifty basketball and football players between the ages of 12 and 18 years old will be examined following informed consent from the children and their legal guardian. Each participant would be measured three times during the year (pre-season, middle-season, and post-season), three times each (before-training, after aerobic warming-up, and after-training) on the Tetrax. Additionally, physical parameters (as height, and weight), anatomical parameters (as leg length), and joint range of movement, would be record.

ELIGIBILITY:
Inclusion Criteria:

* age 12-18 years
* healthy athletes

Exclusion Criteria:

* children with known disturbances in bone, muscle of nervous systems
* children using medications that may cause problems in balance or coordination

Ages: 12 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Thirty basketball and football players between the ages of 12 and 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Posturography measures | Training season
  changes in posturography measures in athletes throughout a training season

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dan Nemet, Kfar Saba, Israel